CLINICAL TRIAL: NCT04689867
Title: Feasibility, Acceptability, and Preliminary Effectiveness of a Cognitive-behavioral Suicide Prevention-focused Intervention Tailored to Adults Diagnosed With Schizophrenia Spectrum Disorders: Aim 1 Open Pilot Trial to Test Modified Treatment and Measurement Prior to Aim 2 RCT (Registered Separately)
Brief Title: Cognitive Behavioral Suicide Prevention for Psychosis: Aim 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lindsay Bornheimer, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00152247; R34MH123609 (NIH)
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Suicide; Psychosis
Keywords: cognitive behavioral therapy; suicide prevention; community mental health
MeSH Terms: conditions — Suicide; Psychotic Disorders; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBSPp (Experimental): Cognitive Behavioral Suicide Prevention for psychosis is a behavioral treatment and will be delivered in 10 weekly individual therapy sessions.
  Interventions: Behavioral: Cognitive Behavioral Suicide Prevention for psychosis CBSPp)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Suicide Prevention for psychosis CBSPp) — Cognitive and behavioral approach to suicide prevention among individuals with psychosis

SUMMARY:
The investigators are modifying and testing the preliminary effectiveness and implementation of a Cognitive Behavioral Suicide Prevention for psychosis (CBSPp) intervention. In this phase of the study, CBSPp will be tested in an initial open trial (n = 10) to examine its feasibility and acceptability. Investigators will recruit clients receiving services at a community mental health setting who have a schizophrenia spectrum disorder and recent suicidal thoughts and behaviors to receive the behavioral intervention for 10-weeks. Providers will be recruited and trained to deliver the intervention. Both clients and providers will be assessed at baseline to test our approach to measurement prior to the Aim 2 RCT (registered separately). Clients will be assessed at three additional timepoints (middle of treatment, end of treatment, and 2 months after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia Spectrum Disorder
* Suicide ideation and/or attempt within 3 months of screening
* Ability to speak and read in English
* 18 to 65 years of age

Exclusion Criteria:

* Requiring emergency care (e.g. imminent plan to harm self) as determined by trained research staff administering the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Inappropriate for behavioral treatment according to own judgment in consultation with a treating clinician CMH
* Impaired capacity (cognitive capacity)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Upload to NIMH Data Archive

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of eight clients consented to participate in the Aim 1 open pilot study and were subsequently scheduled to attend a screening assessment. One individual was not eligible per the screening assessment, and two individuals did not attend the scheduled screening assessment.
  As a result, five individuals were eligible to participate and began treatment.
Groups:
- CBSPp: Cognitive Behavioral Suicide Prevention for psychosis is a behavioral treatment and will be delivered in 10 weekly individual therapy sessions.
  Cognitive Behavioral Suicide Prevention for psychosis CBSPp): Cognitive and behavioral approach to suicide prevention among individuals with psychosis.
  In this open pilot trial, all participants received the treatment.
Period: Overall Study
Arm/Group | CBSPp
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CBSPp
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.66 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Lifetime History of Suicide Attempt [Count of Participants; unit: Participants]
  Yes | 4
  No | 1
Past Week Suicide Attempt [Count of Participants; unit: Participants]
  Yes | 0
  No | 5
Past Week Suicide Ideation [Count of Participants; unit: Participants]
  Yes | 3
  No | 2
Past Week Suicide Plan [Count of Participants; unit: Participants]
  Yes | 3
  No | 2

OUTCOME MEASURES:

1. Primary Outcome: Calgary Depression Rating Scale (CDRS)
Description: A scale to measure depression with scores ranging from 0 to 27 and greater scores indicating greater depression. Item 8 of the scale measures suicide thoughts and behaviors.
Time Frame: baseline, mid-treatment (week 5 of treatment), post-treatment (week 10 of treatment), follow-up (2 months after week 10 of treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSPp
Number analyzed (Participants) | 5
score on a scale
  Baseline | 13.60 (5.73)
  mid-treatment | 9.00 (2.92)
  post-treatment | 11.00 (2.58)
  follow-up | 7.60 (3.65)

2. Primary Outcome: Positive and Negative Symptom Rating Scale (PANSS)
Description: A scale to measure psychosis with item ratings ranging from 1 to 7. There are 3 sub-scales across 30 questions of the full scale: positive symptom scale (score range 7-49), negative symptom scale (score range 7-49), and general symptom scale (score range 16-112). Scores are summed for each of the 3 sub-scales with higher scores indicating greater presence of symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSPp
Number analyzed (Participants) | 5
score on a scale
  Baseline positive sub scale | 20.20 (3.27)
  Baseline negative sub scale | 18.20 (5.89)
  Baseline general sub scale | 42.40 (7.96)
  Mid-treatment positive sub scale | 20.40 (4.16)
  Mid-treatment negative sub scale | 19.00 (7.81)
  Mid-treatment general sub scale | 41.20 (8.53)
  Post-treatment positive sub scale | 20.00 (7.62)
  Post-treatment negative sub scale | 17.75 (6.40)
  Post-treatment general sub scale | 37.50 (10.38)
  Follow-up positive sub scale | 20.80 (7.66)
  Follow-up negative sub scale | 18.00 (8.25)
  Follow-up general sub scale | 43.4 (12.42)

3. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: A scale to measure suicide thoughts and behavior.
  The following are C-SSRS items that have binary responses (yes/no): wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with some intent to act and without specific plan, active suicidal ideation with specific plan and intent, preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal), and suicide death.
  A numerical suicidal ideation score is assigned for the first 5 binary items ranging from 0 (no ideation) to 5 (active ideation with plan and intent)
Time Frame: as for outcome 1
Population: One individual at post-treatment did not complete the assessment with research staff
Measure: Count of Participants; unit: Participants
Arm/Group | CBSPp
Number analyzed (Participants) | 5
Participants
  Baseline suicide ideation: Yes | 3
  Baseline suicide ideation: No | 2
  Baseline suicide plan: Yes | 3
  Baseline suicide plan: No | 2
  Baseline suicide attempt: Yes | 0
  Baseline suicide attempt: No | 5
  Mid-treatment suicide ideation: Yes | 3
  Mid-treatment suicide ideation: No | 2
  Mid-treatment suicide plan: Yes | 4
  Mid-treatment suicide plan: No | 1
  Mid-treatment suicide attempt: Yes | 0
  Mid-treatment suicide attempt: No | 5
  Post-treatment suicide ideation: number analyzed (Participants) | 4
  Post-treatment suicide ideation: Yes | 2
  Post-treatment suicide ideation: No | 2
  Post-treatment suicide plan: number analyzed (Participants) | 4
  Post-treatment suicide plan: Yes | 1
  Post-treatment suicide plan: No | 3
  Post-treatment suicide attempt: number analyzed (Participants) | 4
  Post-treatment suicide attempt: Yes | 0
  Post-treatment suicide attempt: No | 4
  Follow-up suicide ideation: Yes | 3
  Follow-up suicide ideation: No | 2
  Follow-up suicide plan: Yes | 2
  Follow-up suicide plan: No | 3
  Follow-up suicide attempt: Yes | 0
  Follow-up suicide attempt: No | 5

4. Secondary Outcome: Beck Hopelessness Scale
Description: A scale to measure hopelessness using 20 items with binary (true/false) response categories. Scores are summed and range from 0-20, higher scores indicate greater hopelessness is present.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSPp
Number analyzed (Participants) | 5
score on a scale
  Baseline | 12.80 (8.17)
  Mid-treatment | 10.40 (8.76)
  Post-treatment | 12.00 (7.44)
  Follow-up | 9.80 (8.87)

5. Secondary Outcome: The Entrapment Scale
Description: A scale to measure entrapment using 16 items and response categories ranging from 0 to 4. Scores are summed with a range of 0 to 64, and higher scores indicate greater feelings of being entrapped.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSPp
Number analyzed (Participants) | 5
score on a scale
  Baseline | 35.80 (15.61)
  Mid-treatment | 30.40 (21.10)
  Post-treatment | 28.75 (18.39)
  Follow-up | 36.0 (21.09)

6. Secondary Outcome: The Defeat Scale
Description: A scale to measure defeat using 16 items and response categories ranging from 0 to 4. Scores are summed with a range of 0 to 64, higher scores indicate greater feelings of being defeated.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSPp
Number analyzed (Participants) | 5
score on a scale
  Baseline | 43.00 (18.41)
  Mid-treatment | 40.40 (20.62)
  Post-treatment | 39.00 (15.43)
  Follow-up | 41.5 (14.27)

ADVERSE EVENTS:
Time Frame: Adverse event data collected across participant involvement in study (beginning with the eligibility screener and ending after follow-up assessment): Approximately across 5 months per participant
Description: Systematic Assessment of Adverse Events: Routine determination of adverse events through standard assessment at each study timepoints by research staff, project coordinator, or principal investigator.
Arm/Group | CBSPp
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBSPp (N=5)
Anxiety during assessment (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an open pilot trial, therefore no randomization occurred nor comparison between receiving treatment or not. All participants received treatment. The next phase of our study (Aim 2; registered separately) will report on the RCT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT04689867/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT04689867/ICF_001.pdf